CLINICAL TRIAL: NCT02229838
Title: Safety/Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of 0.25 mg, 0.75 mg, 2 mg, 6 mg, and 10 mg BIBB 1464 MS (Tablet) in Healthy Male Subjects, Combined With Preliminary Evaluation of Relative Bioavailability and Effect of Food of the Dose of 0.75 mg or 2 mg or 6 mg (Two-stage Trial Design With Randomised Double Blind Placebo Controlled Rising Dose Phase and Subsequent Randomised, Open Parallel Group Phase)
Brief Title: Safety/Tolerability, Pharmacokinetics, and Pharmacodynamics of BIBB 1464 MS in Healthy Male Subjects, Combined With Preliminary Evaluation of Relative Bioavailability and Effect of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1178.1
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (4):
- BIBB 1464 MS single rising dose fed (Experimental)
  Interventions: Drug: BIBB 1464 MS tablet; Other: Standard dinner
- BIBB 1464 MS tablet fasted (Experimental)
  Interventions: Drug: BIBB 1464 MS tablet
- BIBB 1464 MS solution fasted (Active Comparator)
  Interventions: Drug: BIBB 1464 MS solution
- BIBB 1464 MS placebo (Placebo Comparator)
  Interventions: Drug: BIBB 1464 MS placebo

INTERVENTIONS:
Drug: BIBB 1464 MS tablet
  Arms: BIBB 1464 MS single rising dose fed; BIBB 1464 MS tablet fasted
Drug: BIBB 1464 MS solution
  Arms: BIBB 1464 MS solution fasted
Drug: BIBB 1464 MS placebo
  Arms: BIBB 1464 MS placebo
Other: Standard dinner
  Arms: BIBB 1464 MS single rising dose fed

SUMMARY:
Safety, pharmacodynamics and pharmacokinetics of 0.25, 0.75, 2.0, 6.0, and 10 mg BIBB 1464 p.o once daily in a rising dose group-comparison (placebo controlled, double blind, randomized per dose level).

Relative Bioavailability of 0.75 mg or 2 mg or 6 mg ( tablet vs. solution, intraindividual comparison), preliminary assessment of food effects (interindividual comparison)

Two-stage Trial Design With Randomised Double Blind Placebo Controlled Rising Dose Phase and Subsequent Randomised, Open Parallel Group Phase).

MS (Tablet) in Healthy Male Subjects, Combined With Preliminary Evaluation of Relative Bioavailability and Effect of Food of the Dose of 0.75 mg or 2 mg or 6 mg (Two-stage Trial Design With Randomised Double Blind Placebo Controlled Rising Dose Phase and Subsequent Randomised, Open Parallel Group Phase).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age > 18 and < 55 years
* Broca > - 20% and < + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal (including thyroid) disorder
* Surgery of the gastro-intestinal tract (except appendectomy)
* Disease of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the result of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 month prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or >3 pipes/day)
* Inability to refrain from smoking during the period of the study
* Known alcohol (>60 g/day) or drug abuse
* Blood donation (<=1 month prior to administration)
* Excessive physical activities (<5 days prior to administration)
* Any laboratory value outside the normal range of clinical relevance
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma

Ages: 19 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 1999-07; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Maximum drug plasma concentration (Cmax) | Up to 38 hours after drug administration
Time to reach the maximum concentration of the analyte in plasma (tmax) | Up to 38 hours after drug administration
Total area under the plasma drug concentration-time curve (AUC) | Up to 38 hours after drug administration
Apparent terminal half-life of the analyte in plasma (t1/2) | Up to 38 hours after drug administration
Total plasma clearance divided by the systemic availability factor (CL/f) | Up to 38 hours after drug administration
Dose normalized AUC0-38h ( NAUC0-38h) | Up to 38 h after drug administration
Mean residence time, total (MRTtot) | Up to 38 hours after drug administration
Number of patients with adverse events | Up to 72 hours after last drug administration
Number of patients with clinical significant findings in vital signs | Up to 38 hours after drug administration
Number of patients with clinical significant findings in electrocardiogram (ECG) | Up to 38 hours after drug administration
Number of patients with clinical significant findings in physical examination | Up to 38 hours after drug administration
Investigator assessed tolerability on a 4 point scale | Up to 38 hours after drug administration
Monoepoxysqualene (MES) plasma concentration | Up to 38 hours after drug administration
Amount of drug excreted in urine | Up to 38 h after drug administration